CLINICAL TRIAL: NCT06258369
Title: Gait Initiation and Transition From Double to Single Support in Patients With Unilateral Primary Coxarthrosis Who Have Not Undergone Surgery and Before/After Arthroplasty
Brief Title: Gait Initiation and Transition From Double to Single Support in Patients With Unilateral Primary Coxarthrosis
Acronym: COXAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC-P00122
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary; Coxarthrosis
Keywords: Coxarthrosis; Hip; Arthroplasty; Gait initiation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Patients with coxarthrosis (any stage) without surgery
  Patients with coxarthrosis (any stage) with THP (Total Hip replacement)
  Patients with coxarthrosis (any stage) with RHT (Hip resurfacing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with primary coxarthrosis (any stage). (Other)
  Interventions: Other: Patients with primary coxarthrosis (any stage).
- Patients with primary coxarthrosis (any stage) and operated with Total Hip prosthesis (THP). (Experimental)
  Interventions: Other: Patients with primary coxarthrosis (any stage) and operated with Total Hip Prosthesis (THP).
- Patients with primary coxarthrosis (any stage) and operated with RTH (Hip resurfacing). (Experimental)
  Interventions: Other: Patients with primary coxarthrosis (any stage) and operated with RTH (Hip resurfacing).

INTERVENTIONS:
Other: Patients with primary coxarthrosis (any stage). — Patients who do not undergo surgery will be called specifically for the study to attend a consultation dedicated to gait assessment.
  Arms: Patients with primary coxarthrosis (any stage).
Other: Patients with primary coxarthrosis (any stage) and operated with Total Hip Prosthesis (THP). — Patients scheduled for THP (Total Hip Prosthesis) will be seen at the consultation the day before surgery, in the same hospital as the THP, or at an existing dedicated consultation scheduled for all THP patients. During these scheduled visits, they will be received in the gait analysis laboratory for a gait assessment (V1). Patients will be seen again at 6 months post-operatively for a second gait assessment (V2).
  Arms: Patients with primary coxarthrosis (any stage) and operated with Total Hip prosthesis (THP).
Other: Patients with primary coxarthrosis (any stage) and operated with RTH (Hip resurfacing). — Patients scheduled for RTH (Hip Resurfacing) will be seen at the consultation the day before surgery, in the same hospital as the RTH, or at an existing dedicated consultation scheduled for all RTH patients. During these scheduled visits, they will be received in the gait analysis laboratory for a gait assessment (V1). Patients will be seen again at 6 months post-operatively for a second gait assessment (V2).
  Arms: Patients with primary coxarthrosis (any stage) and operated with RTH (Hip resurfacing).

SUMMARY:
The study consists to evaluate the impact of prosthetic surgery (PTH and RTH) on kinematic and dynamic parameters (joint torques) of the lower limbs during gait initiation in patients with primary coxarthrosis.

Patients included in the study will undergo a three-dimensional gait analysis. Dynamic gait analysis is multidimensional, measuring kinematic parameters (joint amplitudes: ankles, knees, hips, etc.) and dynamic parameters (assessment of joint torque from ankle, knee, hip to lower limb during gait initiation).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 and over
* With primary coxarthrosis (any stage)
* Consulting in the orthopedic departments of participating centers in anticipation of hip surgery (PTH/RTH), or for advice only.
* Written consent signed by the patient
* Affiliation with a social security scheme

Exclusion Criteria:

* Disabling orthopaedic conditions:

Symptomatic contralateral hip/knee disease Symptomatic gonarthrosis or homolateral total knee prosthesis History of surgery on the affected hip History of fracture of the lower limb in the past year History of lower limb sprain in the last 3 months Neurological or degenerative disease

* Pregnant or breast-feeding
* Adults under guardianship, curatorship or safeguard of justice
* Cognitive impairment making it impossible to understand the protocol
* Approach other than Moore posterolateral (for PTH and RTH groups)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2027-08-19 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Amplitude degree of lower limbs articulations | 6 months
Dynamics of limbs joint torques during walking initiation measured in Nm/kg | 6 months

SECONDARY OUTCOMES:
Step length during gait initiation | 6 months
Step width during gait initiation | 6 months
Duration of first step during gait initiation | 6 months
Duration of anticipatory postural adjustment phase during gait initiation | 6 months
Duration of execution phase during gait initiation | 6 months
Measurement of the trajectory during gait initiation | 6 months
Measurement of the speed during gait initiation | 6 months
Measurement of the amplitude of retreat of the center of pressure during gait initiation | 6 months
Severity of coxarthrosis according to the Tönnis classification | 6 Months
  The severity of coxarthrosis is assessed on radiographs according to the Tönnis classification:
  Grade Radiographic features 0 - No signs of osteoarthritis
  1. - Slight narrowing of joint space
     * Slight lipping at joint margin
     * Slight sclerosis of the femoral head or acetabulum
  2. - Small cysts in the femoral head or acetabulum
     * Increasing narrowing of joint space
     * Moderate loss of sphericity of the femoral head
  3. - Large cysts
     * Severe narrowing or obliteration of joint space
     * Severe deformity of the femoral head
     * Avascular necrosis
HHS (Harris Hip Score) | 6 months
  The functional score consists of 10 items out of 100 points (best score = 100 points) assessing function, pain and mobility
PMA (Postel Merle d'Aubigné) score | 6 months
  Score on 3 items (pain, mobility and walking) rated on 18 points (18 = excellent results, 0 = worst result)
Devane score | 6 months
  Activity score with 5 possibilities (1 = sedentary work and 5 = power work, competitive sport)
UCLA (University of California Los Angeles) score | 6 months
  Activity score comprising 10 possibilities and assessing the intensity of physical activity (1= inactive or dependent patient, 10 = regular practice of high-impact sports)
Vellas unipodal weight-bearing test | 6 months
  This test consists in asking the patient to balance for as long as possible. A time of more than 30 seconds indicated a very low risk of falls. A time of less than 5 seconds indicates a very high risk of falls.
Pelvic incidence | 6 months
  Pelvic incidence is a constant morphologic parameter that describes the "pelvic size" based on the angular relation between femoral heads and sacral plate for any given person
Sacral slope angle | 6 months
  Spatial orientation of the pelvis in the sagittal plane is assessed by the sacral slope
Pelvic tilt angle | 6 months
  Pelvic tilt is a position-dependent parameter defined as the angle created by a line running from the sacral endplate midpoint to the center of the bifemoral heads and the vertical axis.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MARTINOT, MD, Study Director — Hôpital Saint Philibert, GHICL
Locations (2):
- France (2):
  - CHU de Lille, Lille
  - Hôpital Saint-Philibert (GHICL), Lomme